CLINICAL TRIAL: NCT05826158
Title: 18F-mFBG LAFOV PET/CT Compared to 123I-mIBG Scintigraphy SPECT/CT for Evaluation of Children With Neuroblastoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Lise Borgwardt, Senior Consultant Ph.D., Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: j. nr. H-21009982_v3
Record Dates: First submitted 2023-04-11; First posted 2023-04-24 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Neuroblastoma
Keywords: 18F-mFBG; meta-fluorobenzylguanidine; Large Axial Field of View PET/CT, LAFOV PET/CT; Total body PET/CT
MeSH Terms: conditions — Neuroblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Children with Neuroblastoma (Other)
  Interventions: Diagnostic Test: 18FmFBG imaging on the Large Field of View PET/CT (Total body PET/CT)

INTERVENTIONS:
Diagnostic Test: 18FmFBG imaging on the Large Field of View PET/CT (Total body PET/CT) — 18F-mFBG imaging on the Large Field of View PET/CT (Total body PET/CT)

SUMMARY:
This is a study evaluating the positron-emitting radiopharmaceutical 18F-mFBG compared to 123I-mIBG scintigraphy for imaging of neuroblastoma

DETAILED DESCRIPTION:
This is a prospective study designed to assess the use of 18F-mFBG PET imaging compared to 123I-mIBG scintigraphy in subjects with known or presumed neuroblastoma. Eligible participants will have either histopathologically established diagnosis of neuroblastoma or a presumed diagnosis based on signs, symptoms, physical examination, imaging findings, and laboratory and genetic test results.

Subjects will only be administered 18F-mFBG if they have undergone or are scheduled to undergo a 123I-mIBG within +/- 7 days of the date of the 18F-mFBG scan. Subjects should not have received any chemotherapy, immunotherapy or radiotherapy between the clinical and 18F-mFBG imaging studies.

18F-mFBG PET studies will be evaluated by 2 independent teams of blinded readers: a nuclear medicine physician and a radiologist, both specialized in pediatric nuclear medicine co-reading side-by side.

The clinical 123I-mIBG is also evaluated by 2 independent teams of blinded readers: a nuclear medicine physician and a radiologist, both specialized in pediatric nuclear medicine co-reading side-by side.

Blinded readers will record whether findings on 18F-mFBG and 123I-mIBG scans are consistent with neuroblastoma.

Subject-level diagnostic performance will be assessed on the basis of differencies in lesion-counting between the blinded 18F-mFBG scan interpretation and the 123I-mIBG scan. In case of discrepancy, independently assessed by an Expert Panel.

ELIGIBILITY:
Inclusion Criteria:

1. An established diagnosis of neuroblastoma based on unequivocal histopathology from tissue obtained at any time prior to enrolment in the trial; OR b) A presumed diagnosis of neuroblastoma based on signs, symptoms, physical examination, imaging findings, and laboratory and genetic test results, including individuals in whom therapy has already been empirically initiated.
2. The subject has undergone or is scheduled to undergo evaluation of neuroblastoma disease status, including 123I-mIBG +/- 7 days to the date of 18F-mFBG imaging, with no therapy between such evaluation.
3. Ability of subject or subject's legal guardian to understand and sign a written informed consent document.

   -

   Exclusion Criteria:

1. Pregnancy

-

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-06-06 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
18F-mFBG PET Scan identification of Neuroblastoma on the LAFOV PET/CT | 60 minutes
  Pathological 18F-mFBG uptake when imaging after 60 minutes with LAFOV PET/CT

SECONDARY OUTCOMES:
Comparison of 18F-mFBG with Clinical 123I-mIBG imaging | 7 days apart
  Pathological uptake on 18F-mFBG will be compared with pathological uptake on 123I-mIBG, lesions based comparison

CONTACTS AND LOCATIONS:
Overall Officials: Lise Borgwardt, MD, PhD., Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen University Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No